CLINICAL TRIAL: NCT00000530
Title: Raynaud's Treatment Study (RTS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: 73
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2004-08

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Raynaud's Disease; Vascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Raynaud Disease; Vascular Diseases | interventions — Nifedipine; Biofeedback, Psychology; Neurofeedback

INTERVENTIONS:
Drug: nifedipine
Behavioral: biofeedback (psychology)
Procedure: electromyography

SUMMARY:
To determine the relative efficacy of usual medical care and a course of treatment by thermal biofeedback in reducing vasospastic attacks characteristic of Raynaud's syndrome. Also, to confirm the frequency and severity of attacks, examine the role of psychophysiological factors in precipitating attacks, and assess the influence of treatment on health quality of life.

DETAILED DESCRIPTION:
BACKGROUND:

Primary Raynaud's phenomenon is a peripheral vascular disorder resulting in vasospastic attacks provoked by cold and/or emotional stress. Attacks most often occur in the fingers, but may occur in other extremities as well.

DESIGN NARRATIVE:

Randomized. Patients were assigned to one of four treatment groups: slow release Nifedipine, a calcium channel blocker; pill placebo; temperature biofeedback; or electromyograph biofeedback from the frontalis muscle. The primary endpoint was reduction in number of vasospastic attacks. Other endpoints included: other measures of Raynaud's attacks including frequency, severity, duration, response to laboratory-based cold challenge, and quality of life.

ELIGIBILITY:
Men and women with documented primary or secondary Raynaud's syndrome.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1992-09; Study Completion 1998-06

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Thompson — Clinical Trials & Surveys Corp (C-TASC)

REFERENCES:
- [Background] Jennings JR, Maricq HR, Canner J, Thompson B, Freedman RR, Wise R, Kaufmann PG. A thermal vascular test for distinguishing between patients with Raynaud's phenomenon and healthy controls. Raynaud's Treatment Study Investigators. Health Psychol. 1999 Jul;18(4):421-6. doi: 10.1037//0278-6133.18.4.421. PMID 10431945
- [Background] Comparison of sustained-release nifedipine and temperature biofeedback for treatment of primary Raynaud phenomenon. Results from a randomized clinical trial with 1-year follow-up. Arch Intern Med. 2000 Apr 24;160(8):1101-8. doi: 10.1001/archinte.160.8.1101. PMID 10789602
- [Background] Brown KM, Middaugh SJ, Haythornthwaite JA, Bielory L. The effects of stress, anxiety, and outdoor temperature on the frequency and severity of Raynaud's attacks: the Raynaud's Treatment Study. J Behav Med. 2001 Apr;24(2):137-53. doi: 10.1023/a:1010758530555. PMID 11392916
- [Background] Maricq HR, Jennings JR, Valter I, Frederick M, Thompson B, Smith EA, Hill R; Raynaud's Treatment Study Investigators. Evaluation of treatment efficacy of Raynaud phenomenon by digital blood pressure response to cooling. Raynaud's Treatment Study Investigators. Vasc Med. 2000;5(3):135-40. doi: 10.1177/1358836X0000500302. PMID 11104295
- [Background] Middaugh SJ, Haythornthwaite JA, Thompson B, Hill R, Brown KM, Freedman RR, Attanasio V, Jacob RG, Scheier M, Smith EA. The Raynaud's Treatment Study: biofeedback protocols and acquisition of temperature biofeedback skills. Appl Psychophysiol Biofeedback. 2001 Dec;26(4):251-78. doi: 10.1023/a:1013182519331. PMID 11802676
- [Background] Thompson B, Geller NL, Hunsberger S, Frederick M, Hill R, Jacob RG, Smith EA, Kaufmann P, Freedman RR, Wigley FM, Bielory L. Behavioral and pharmacologic interventions: the Raynaud's Treatment Study. Control Clin Trials. 1999 Feb;20(1):52-63. doi: 10.1016/s0197-2456(98)00046-4. PMID 10027500
- Available data/document: Individual Participant Data Set: RTS — http://biolincc.nhlbi.nih.gov/studies/rts/ — NHLBI provides controlled access to IPD through BioLINCC. Access requires registration, evidence of local IRB approval or certification of exemption from IRB review, and completion of a data use agreement.
- Available data/document: Study Protocol — http://biolincc.nhlbi.nih.gov/studies/rts/
- Available data/document: Study Forms — http://biolincc.nhlbi.nih.gov/studies/rts/